CLINICAL TRIAL: NCT02418234
Title: Frequency and Abundance of T790M Mutation on Circulating Tumor DNA in Patients With Non-small Cell Lung Cancer After Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors Treatment Failure: a Perspective Observational Study
Brief Title: T790M Mutation on ctDNA in Patients With NSCLC After EGFR-TKI Failure
Status: Completed | Type: Observational
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: HZFH CA15-02
Record Dates: First submitted 2015-04-03; First posted 2015-04-16 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-01

CONDITIONS: Non-small Cell Lung Cancer Stage III; Non-Small-Cell Lung Cancer Metastatic
Keywords: Non-small Cell Lung Cancer; circulating tumor DNA; T790M; amplification refractory mutation system; digital droplet PCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: mutation detection
Other: ARMS and ddPCR
Genetic: ctDNA analysis

SUMMARY:
The purpose of this study is to compare the frequency and abundance of T790M mutation among the different Clinical modes of EGFR-TKI failure.

DETAILED DESCRIPTION:
An observational, non-interventional, multi-central study of comparison of the frequency and abundance of T790M mutation using both amplification refractory mutation system (ARMS) and digital droplet PCR (ddPCR) methods among the different Clinical modes of non-small cell lung cancer (NSCLC) patients with epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) failure

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB/IV NSCLC.
* Investigator confirmed progression according RECIST 1.1 during EGFR-TKI treatment within 28 days of the enrollment
* Activating mutation (G719A/C/S; Exon 19 insertion/deletion; L858R; L861Q) in the EGFR gene or have had at least partial response with EGFR TKI lasting ≥ 6 months
* Patient must be able to comply with the protocol

Exclusion Criteria:

* Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 defined disease progression for more than 28 days while on previous EGFR-TKI treatment.
* Patient has been treated with any investigational agent for any indication within 4 weeks of study treatment.
* Histologically confirmed small cell lung cancer or other metastatic tumors
* Patient with no histologic or cytological diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non small cell lung cancer (NSCLC) after EGFR-TKI failure
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

RESULTS

PARTICIPANT FLOW:
Groups:
- TKI-PD: Patients with advanced or recurrent NSCLC who had progressed during EGFR-TKIs treatment
Period: Overall Study
Arm/Group | TKI-PD
Started | 314
Completed | 314
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- TKI-PD: Patients with advanced or recurrent NSCLC patients had progressed during EGFR-TKIs treatment
Arm/Group | TKI-PD
Number analyzed (Participants) | 314
Age, Continuous [Median (Full Range); unit: years] | 63 [32 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177
  Male | 137
Region of Enrollment [Number; unit: participants]
  China | 314
Stage [Number; unit: participants] — Each patient was staged according to NCCN guidelines (2015. v6) at the time of enrollment. Generally, Stage IV showed worse prognosis.
  participants
    IIIA | 54
    IIIB | 21
    IV | 239

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With T790M Mutation Detected by Amplification Refractory Mutation System (ARMS) Assay
Description: The investigators will describe the number of T790M mutation on ctDNA detected by ARMS assay in patients with non-small cell lung cancer (NSCLC) resistant to tyrosine kinase inhibitors (TKIs).
Time Frame: up to 2 years
Measure: Number; unit: participants
Arm/Group | TKI-PD
Number analyzed (Participants) | 314
participants | 97

2. Primary Outcome: Abundance of T790M Mutation Detected by Digital Droplet PCR (ddPCR) Assay in Each Individual Patient
Description: The investigators will describe the abundance of T790M mutation on ctDNA detected by ddPCR assay in patients with NSCLC resistant to TKIs.
Time Frame: up to 2 years
Measure: Median (Full Range); unit: percentage of total ctDNA
Arm/Group | TKI-PD
Number analyzed (Participants) | 314
percentage of total ctDNA | 0 [0 to 70.3]

3. Secondary Outcome: Number of T790M Mutation by ARMS and ddPCR Assays in Each Different Clinical Modes of TKI Failure
Description: The investigators will describe the number of participants with T790M mutation in each different clinical mode of TKI failure by ARMS and ddPCR, and employ chi-square test to analyze the distribution of T790M mutation by ARMS and ddPCR in patients among the different Clinical modes of TKI failure.
Time Frame: up to 2 years
Measure: Number; unit: participants
Groups:
- Chest Limited: Chest limited was defined as progressive disease (PD) in lung/pleura tissue and lymph nodes limited in chest, and no evidence of progression beyond the chest was identified.
- Brain Limited: Brain limited was defined as a PD in original site or a new site of metastatic disease in brain, with no evidence of extracranial progression.
- Other Sites Failures: Other sites failures were defined as PD lesions in other distant site, or multiple sites including chest or intracranial.
Arm/Group | Chest Limited | Brain Limited | Other Sites Failures
Number analyzed (Participants) | 196 | 34 | 84
participants
  T790M positive by ARMS | 49 | 2 | 46
  T790M positive by ddPCR | 78 | 7 | 62
Statistical Analysis 1: Comparison: Chest Limited vs Brain Limited vs Other Sites Failures; Test type: Superiority or Other; p < 0.05, Chi-squared

4. Secondary Outcome: Differences of T790M Mutation by ddPCR Among the Different Clinical Modes of TKI Failure
Description: The investigators will employ Analysis of Variance (ANOVA) method to analyze the differences of T790M mutation by ddPCR in patients among the different Clinical modes of TKI failure.
Time Frame: up to 2 years
Measure: Median (Full Range); unit: percentage of total ctDNA
Arm/Group | Chest Limited | Brain Limited | Other Sites Failures
Number analyzed (Participants) | 196 | 34 | 84
percentage of total ctDNA | 0 [0 to 34.61] | 0 [0 to 13.07] | 0.56 [0 to 70.3]
Statistical Analysis 1: Comparison: Chest Limited vs Brain Limited vs Other Sites Failures; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | TKI-PD
Serious Adverse Events (participants affected / at risk) | 0/314
Other Adverse Events (participants affected / at risk) | 0/314

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No